CLINICAL TRIAL: NCT04791306
Title: Impact of a 4 Months Training Intervention on Exercise-induced Changes of Heart Health-related Epigenetic Markers in Healthy, Sedentary Individuals
Brief Title: Impact of 4 Months of Exercise Changes of Heart Health-related Epigenetic Markers in Healthy, Sedentary Individuals
Acronym: miR-4-heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Collaborators: Ludwig Boltzmann Institute for Digital Health and Prevention (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Prim. Univ.Prof.Dr.Dr. Josef Niebauer, MBA, Paracelsus Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UISM-13
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Training (Experimental): All participants should increase their physical activity level to at least 150 min per week, guided with once a week supervised in-house training as well as an application for planning and documentation for home-based physical activity
  Interventions: Other: supervised exercise training; Other: home-based exercise training

INTERVENTIONS:
Other: supervised exercise training — Participates perform once a week for 4 months an in-house supervised endurance and strength training.
Other: home-based exercise training — Participants are provided with an application for planning and documentation of their physical activity, together with an expert participants plan their physical activities for their home-based training to reach at least 150 min physical activity per week.

SUMMARY:
We aim to analyze the impact of a single acute exercise intervention (ergometry) on the expression pattern of specific heart health related miRNAs in healthy, previously sedentary participants, and how this pattern will be changed after 4 months of increasing the weekly physical activity >150 minutes.

DETAILED DESCRIPTION:
Exercise induced changes in heat health related miRNA expression pattern are analyzed in plasma samples collected at rest and immediately after the completion of an all-out ergo spirometry test, conducted during the baseline examination. Additionally participants will perform a pulse wave analysis to evaluate their arterial stiffness, a bioimpedanzanalysis to evaluate their body composition, blood lipids will be measured as well as their exercise capacity.

After the baseline examination, all participants will perform once per week a supervised endurance and strength training at our facility. In addition, the participants will be provided with a digital application for planning and documentation of their home based physical activity. Together with an expert, they plan their weekly physical activities so that they reach 150 min of physical activity each week over a period of 4 months.

After this training/exercise intervention all participants will perform all measurements from the baseline examination again.

ELIGIBILITY:
Inclusion Criteria:

* <150min physical activity per week
* >18 years of age
* male and female
* signed inform consents

Exclusion Criteria:

* acute or chronic cardiovascular diseases, exempt arterial hypertension (systolic blood pressure >140 mmHg and diastolic blood pressure >90 mmHg in untreated and medical treated subjects)
* acute or chronic lung disease
* Alcohol (>30g/day) or drug abuse
* Adipositas grad 2 (BMI >35kg/m²)
* Orthopedic limitations to exercise capacity
* pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
miRNA expression response to acute all-out exercise (ergometry) | Baseline
  expression change of miRNA due to all-out ergometry at baseline
Change from baseline miRNA expression at 4 months | after 4 months of exercise intervention
  4 months of exercise intervention in healthy previously sedentary participants leads to exercise-induced changes in the cardio protective miRNA expression profiles
Change from baseline in miRNA expression response to acute all-out exercise (ergometry) at 4 months | after 4 months of exercise intervention
  4 months of exercise intervention in healthy previously sedentary participants leads to a change in the acute exercise response (all-out ergometry).

SECONDARY OUTCOMES:
Heart rate | Before and after 4 months of exercise intervention
  Heart rate will be measured by graded exercise testing on cycle ergometer.
blood lipides | Before and after 4 months of exercise intervention
  blood lipides will be measured before and after intervention
arterial stiffness | Before and after 4 months of exercise intervention
  arterial stiffness will be measured before and after intervention
body composition | Before and after 4 months of exercise intervention
  body composition will be measured before and after intervention
exercise capacity | Before and after 4 months of exercise intervention
  exercise capacity will be measured by graded exercise testing on cycle ergometer.
body weight | Before and after 4 months of exercise intervention
  body weight will be measured before and after intervention
digital application | 4 months of exercise intervention
  user feedback and user experience will be evaluated after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Josef Niebauer, MD PhD MBA, Principal Investigator — Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University
Locations (1):
- Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University, Salzburg, Austria